CLINICAL TRIAL: NCT01921881
Title: Does the Natural Medicinal Plant St John's Wort Affect the Glucose Tolerance in Healthy Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tore B. Stage, MSc Pharm, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AKF-385
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes
Keywords: Glucose tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hypericum extract LI 160

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- St John's wort (Experimental): Subjects will undergo 3 oral glucose tolerance tests:
  1. Without taking any St John's wort
  2. After 3 weeks pretreatment with St John's wort
  3. Minimum 6 weeks after last St John's wort ingestion
  Interventions: Other: St John's wort

INTERVENTIONS:
Other: St John's wort

SUMMARY:
The goal of the study is to examine if healthy individuals that ingest St John's wort will have a significantly difference in glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Males
* Fasting plasma-glucose < 7.0 mmol/L
* Glycosylated haemoglobin A1c within reference or clinically insignificant deviation hereof
* Body mass index < 30 kg/m^2

Exclusion Criteria:

* Hypersensitivity to St John's wort
* Chronical or daily alcohol abuse
* Known liver disease
* Ingestion of drugs requiring prescription, except locally acting drugs

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Glucose area under curve (AUC) 0-2 hours | Glucose concentration 0, 15, 30, 45, 60, 90 and 120 after glucose ingestion
  At time=0, the subjects will ingest 75g glucose. Plasma glucose will be measured at 0, 15, 30, 45, 60, 90 and 120 minutes after glucose ingestion.

SECONDARY OUTCOMES:
St John's wort pharmacokinetics | At time=0
  At time=0, the concentration of active components hypericin and hyperforin will be measured.
Other metabolic markers | At time points, 0, 15, 30, 45, 60, 90, 120 minutes after glucose ingestion
  C-peptide and serum insulin will also be measured during the oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brøsem, Professor, MD, Study Director — University of Southern Denmark; Per Damkier, MD PhD, Principal Investigator — University of Southern Denmark; Tore B. Stage, MSc Pharm, Principal Investigator — University of Southern Denmark
Locations (1):
- Department of Clinical Pharmacology, Institute of Public Health, University of Southern Denmark, Odense C, Denmark